CLINICAL TRIAL: NCT00401856
Title: A Randomised, Double-blinded, Placebo-controlled Trial Using Cardiovascular Magnetic Resonance (CMR) Scanning to Assess Remodelling and Regression of Fibrosis in Cardiomyopathy With Eplerenone
Brief Title: CMR to Assess Fibrosis in Cardiomyopathy Using Eplerenone
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Royal Brompton & Harefield NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2004CD006B; Eudract 2004-002494-23
Record Dates: First submitted 2006-11-20; First posted 2006-11-22 (Estimated); Last update posted 2021-09-21 (Actual); Status verified 2021-09

CONDITIONS: Cardiomyopathy
Keywords: Cardiomyopathy; Fibrosis; Magnetic-Resonance; Eplerenone
MeSH Terms: conditions — Cardiomyopathies; Fibrosis | interventions — Eplerenone

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- 1 (Experimental): This arm will receive eplerenone
  Interventions: Drug: Eplerenone
- 2 (Placebo Comparator): This group will receive the placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Eplerenone — 50mg oral route
  Arms: 1
Drug: Placebo — Placebo is identical to eplerenone but the active ingredient is absent
  Arms: 2

SUMMARY:
The aim of this study is to determine if therapy with the aldosterone antagonist, Eplerenone, is associated with improved remodeling of the left ventricle in patients with cardiomyopathy. We will determine if any benefit to cardiac remodeling is associated with improved clinical outcomes, including improved exercise capacity and reduced incidence of major adverse cardiac events such as death, hospitalization for heart-failure, serious heart rhythm disturbances and transplantation.

The null hypothesis is that therapy with Eplerenone over 12 months is associated with an improvement in cardiopulmonary exercise capacity and furthermore that treatment is associated with improved clinical outcomes.

In order to test this hypothesis we will study stable patients on optimal drug therapy with documented cardiomyopathy using a trial design where therapy will be randomized, double-blinded and placebo-controlled. This will reduce the likelihood of any 'researcher bias'. Patients will be recruited from the Heart-failure Service at the Royal Brompton Hospital.

DETAILED DESCRIPTION:
Our aim is to recruit 140 patients (based on statistical power calculation in). These patients will be recruited from the cardiology clinics at The Royal Brompton Hospital as well as from a database of patients who have previously undergone imaging.

The study will be a double-blinded, placebo-controlled randomized study. The recruited patients would have had an established diagnosis of cardiomyopathy as documented by the history, examination and characteristic echocardiographic + ECG findings. The patients would also have had a CMR scan demonstrating late gadolinium hyperenhancement previously. These patients will have been established on maximally tolerated doses of standard drugs used in the treatment of cardiomyopathy (including ACE inhibitors and beta blockers as appropriate) and the doses of these drugs would have remained unchanged in the 2 months preceding enrollment to the trial. Patients would be randomized to receive a maximal dose of 50mg eplerenone or placebo. The study dose of Eplerenone to be used will be initially 25mg once daily (one tablet). After 4 weeks, provided it has been well tolerated with no problems the dose will be increased to the usual maintenance dose of 50mg once daily (two tablets). For patients receiving placebo, the number of tablets received will match the Eplerenone group at the same time points.

Baseline tests will include CMR evaluation of ventricular function using a magnetic field strength of 1.5 Tesla (T). The initial scan will assess ventricular size and function and LV mass. Blood tests will be taken prior to the scan (at the time of intravenous cannulation) for urea and electrolytes, liver function, cytokines, and collagen markers. In addition, echocardiograms, 24 hour Holter monitors will be fitted and metabolic exercise tests (MVO2) will be performed as part of the cardiac assessment at baseline, 6 and 12 months.

The findings of the initial scans and tests will be correlated with base line parameters and also prospectively compared with the occurrence of events over 6 and 12 month time periods. During the follow up period all events including death, cardiac arrest, cardiac transplantation, arrhythmic events, implantation of implantable cardiac defibrillators/biventricular pacemakers, NYHA classification, escalation of treatment and hospitalization will be recorded. There will be regular clinical reviews at 1 week, 2 weeks, 4 weeks and then at 3, 6, 9 and 12 months during the study period at which point blood tests will be taken including a check of renal function to look for evidence of hyperkalaemia and renal failure which may be a result of treatment with eplerenone. Other reported adverse effects and any withdrawals from the trial as a direct result of these effects will also be recorded. After the treatment/placebo has been stopped we will contact all patients within one week by telephone to ensure that there has been no deterioration in symptoms and will review all patients within four weeks for a post-treatment follow up visit to monitor their blood-pressure, kidney function and ensure that there has been no evidence of problems.

Patients will also be asked to complete a Minnesota Living with Heart Failure (MLWHF) Questionnaire at baseline visit and again during the 6 and 12 month visits.

It is hoped that the study will reveal that patients with cardiomyopathy who are treated with eplerenone will have evidence of regression of fibrosis with a concomitant improvement in diastolic function as demonstrated by CMR scanning, as well as in clinical outcomes by Holter and metabolic exercise testing and markers of collagen turnover.

ELIGIBILITY:
Inclusion Criteria:

* Stable patients with an established diagnosis of cardiomyopathy as assessed by history, examination and typical ECG/Echo findings who are on maximally tolerated doses of appropriate drugs with no changes being made to the prescription in the 2 months preceding the start of the trial.

Exclusion Criteria:

* Patients already established on treatment with an aldosterone antagonist
* Patients with contraindications to eplerenone (hyperkalaemia, renal failure)
* Critically ill patients requiring respiratory and/or circulatory support
* Pacemaker or ICD
* Implanted ferromagnetic cerebrovascular clips
* Pregnant women (precautionary only)
* Intolerance of confined spaces
* Inability to lie supine for 60 minutes
* Unwilling or unable to give written informed consent
* Atrial fibrillation or ventricular bigemini.
* Any contraindication to CMR.
* Recent MI
* HCM patients who have received surgical/alcohol ablation treatment

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2007-12; Primary Completion 2013-04-02 (Actual); Study Completion 2013-04-02 (Actual)

PRIMARY OUTCOMES:
Improvement in MVO2 | 6 months

SECONDARY OUTCOMES:
Reduction in major adverse cardiovascular events | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Sanjay Prasad, MD, MRCP, Principal Investigator — Royal Brompton & Harefield NHS Foundation Trust
Locations (1):
- Royal Brompton & Harefield NHS Trust, London, United Kingdom